CLINICAL TRIAL: NCT00572780
Title: Can CT Enteroclysis Predict the Response to Therapy and Outcome in Patient With Crohn's Disease
Brief Title: Can CT Enteroclysis Predict the Outcome of Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 070759
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; CT Enteroclysis
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CTE with CD: Crohn's disease patients who underwent a CT enteroclysis as part of their clinical evaluation for symptomatic Crohn's disease.

SUMMARY:
Specific CT Enteroclysis findings with or without other clinical and laboratory variables, can identify Crohn's disease patients who will response to medical therapy versus those who will either fail and require surgery or have uncontrolled disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease with CT Enteroclysis during symptomatic treatment

Exclusion Criteria:

* Crohn's disease subjects who have had a follow-up less than 1 year, without surgery
* Crohn's disease subjects that were later diagnosed with a bowel malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease patients that have had a CT Enteroclysis as part of their clinical evaluation for symptomatic Crohn's disease will be eligible. Subjects who were later diagnosied with bowel malignancy and subjects with a period of follow-up of less than 1 year(without surgery) will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Chiorean, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States